CLINICAL TRIAL: NCT04860245
Title: Risks and Outcomes Among COVID-19 Patients Admitted to Assiut University Hospitals.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Moustafa, Resident at chest department Assiut university, Assiut University
Other Study IDs: Risks and Outcomes ofCOVID-
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess risks and outcomes among COVID-19 patients admitted to Assiut University Hospitals.

DETAILED DESCRIPTION:
Corona Virus comprises a large group of viruses, that are common in human beings as well animals. There are seven different strains of corona virus, one of them is SARS-COV-2 (the novel coronavirus that causes coronavirus disease 2019, COVID-19) [1].

On 11th March 2020. The World Health Organization declared the international spread of COVID-19 considering it a global pandemic. On 3rd July 2020. WHO declared the total number of confirmed cases of COVID-19 patients is 10,720,450 and number of deaths is 517,340 cases worldwide while in Egypt number of confirmed cases is 71,299 and number of deaths is 3,120 [2].

The largest disparity found was by age. People who were 80 or older were seventy times more likely to die than those under 40. Higher in males than females. Higher in those living in deprived area than those living in the least deprived and higher in Black, Asian and Minority Ethnic groups than in White ethnic groups [3].

It was found that Demographic Characteristics, underlying health state and clinical presentation affect outcome of COVID-19 patients. For example, incidence highest among people aged > 80 years. Hospitalization is six times higher among patients with reported underlying comorbidity (45.4%) than those without reported underlying comorbidity (7.6%). Deaths were 12 times higher in patients with reported underlying comorbidity (19.5%) compared to those without underlying comorbidity (1.6%) [4,5].

Human to human transmission occurs via droplets, contaminated hands or surfaces with Incubation Period 2-14 days after exposure to virus. clinical presentation include: fever, cough, shortness of breath, new loss of taste and smell, body ache, headache, sore throat and diarrhea [6].

Real time PCR used as diagnostic tool for COVID-19, other laboratory findings include leukopenia, lymphopenia, elevated CRP, elevated D-Dimer, high cytokine levels (IL-2R, IL-6, IL-10, and TNF-α), and high lactate dehydrogenase level were significantly associated with severe COVID-19 on admission [7][8].

Computed Tomography (CT Chest) used for assessment severity of lung affection and follow up. Typical CT findings include Ground Glass Opacities: bilateral, subpleural and peripheral, crazy paving appearance (GGO and inter-/intra-lobular septal thickening), Air space consolidation and bronchovascular thickenings [9].

The main therapies used in treatment include Home Isolation, drugs: antibiotic, antiviral, corticosteroids, multivitamins and anticoagulants, O2 therapy, non invasive intervention e.g.: CPAP and invasive intervention e.g.: Mechanical Ventilation. Outcome of patients depend on several factors e.g.: comorbidities, previous lung state, early diagnosis and start of treatment [10].

ELIGIBILITY:
Inclusion Criteria:

- Cases aged 18 years and over. Cases diagnosed as COVID-19 by radiology or with positive PCR. Cases admitted to Assiut University Hospitals.

Exclusion Criteria:

* Cases less than 18 years old. Cases diagnosed as COVID-19 and discharged from emergency department for Home Isolation. Cases express a dissent from the use of their data in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases aged 18 years and over. Cases diagnosed as COVID-19 by radiology or with positive PCR. Cases admitted to Assiut University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
relation between age and INFECTION WITH COVID19 mortality rate of covid19 | baseline
  ANALYSIS AGE OF PEOPLE GET INFECTED WITH COVID 19 AND MORTALITY RATE

CONTACTS AND LOCATIONS:
Overall Officials: Maha Kamel Ghanem, professor, Study Director — Assiut University; hoda A. makhlouf, professor, Study Director — Assiut University; Ali A. hassan, professor, Study Director — Assiut University; Asmaa M. soliman, assistant prof, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Lu Xuefong, Gong Wei, Wang Li, Li Liang, Xie Baojun. Clinical features and high resolution CT imaging findings of Preliminary diagnosis novel coronavirus pneumonia. Chin J Radiol 2020,54.
- [Background] Zhai P, Ding Y, Wu X, Long J, Zhong Y, Li Y. The epidemiology, diagnosis and treatment of COVID-19. Int J Antimicrob Agents. 2020 May;55(5):105955. doi: 10.1016/j.ijantimicag.2020.105955. Epub 2020 Mar 28. PMID 32234468
- [Background] Li X, Xu S, Yu M, Wang K, Tao Y, Zhou Y, Shi J, Zhou M, Wu B, Yang Z, Zhang C, Yue J, Zhang Z, Renz H, Liu X, Xie J, Xie M, Zhao J. Risk factors for severity and mortality in adult COVID-19 inpatients in Wuhan. J Allergy Clin Immunol. 2020 Jul;146(1):110-118. doi: 10.1016/j.jaci.2020.04.006. Epub 2020 Apr 12. PMID 32294485
- [Background] CDC COVID-19 Response Team. Severe Outcomes Among Patients with Coronavirus Disease 2019 (COVID-19) - United States, February 12-March 16, 2020. MMWR Morb Mortal Wkly Rep. 2020 Mar 27;69(12):343-346. doi: 10.15585/mmwr.mm6912e2. PMID 32214079
- [Background] Garg S, Kim L, Whitaker M, O'Halloran A, Cummings C, Holstein R, Prill M, Chai SJ, Kirley PD, Alden NB, Kawasaki B, Yousey-Hindes K, Niccolai L, Anderson EJ, Openo KP, Weigel A, Monroe ML, Ryan P, Henderson J, Kim S, Como-Sabetti K, Lynfield R, Sosin D, Torres S, Muse A, Bennett NM, Billing L, Sutton M, West N, Schaffner W, Talbot HK, Aquino C, George A, Budd A, Brammer L, Langley G, Hall AJ, Fry A. Hospitalization Rates and Characteristics of Patients Hospitalized with Laboratory-Confirmed Coronavirus Disease 2019 - COVID-NET, 14 States, March 1-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):458-464. doi: 10.15585/mmwr.mm6915e3. PMID 32298251
- See also: World Health Organization Coronavirus Disease (COVID-19) Dashboard. — https://www.who.int/emergencies/diseases/novel-coronavirus-2019?gclid=CjwKCAjwrvv3BRAJEiwAhwOdM4ERWNr-IPeHEBomMmypfjCdEH9uvwRimUMhvR0N0Om8-6CBmqTJsRoCojUQAvD_BwE